CLINICAL TRIAL: NCT06559891
Title: A Pivotal, Prospective, Multicenter, 2:1 Randomized, Double Blind, Controlled, Study Comparing the THerapeutic IntravasculaR Ultrasound (TIVUS™) REnal Denervation System Versus Sham for the Adjunctive Treatment of Hypertension (The THRIVE Study)
Brief Title: THRIVE- THerapeutic IntravasculaR Ultrasound (TIVUS™) REnal Denervation System Versus Sham for the Adjunctive Treatment of Hypertension
Acronym: THRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SoniVie Inc. (Industry)
Collaborators: NAMSA (Other); European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CLNS07-001
Record Dates: First submitted 2024-07-24; First posted 2024-08-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: 2:1 randomization will be used to assign subjects to treatment (RDN) or control (sham). Randomization will occur immediately after the renal angiogram.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The subjects and all study personnel taking follow-up blood pressure measurements will be blinded to the randomization up to 6 months post-randomization. Subjects will complete a blinding assessment prior to hospital discharge, at 2M and 6M FU. Study unblinding will occur at 6-months FU.
  ABPM measurements will be sent to an independent core lab for data cleaning and analysis and will be blinded to the randomization assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- TIVUS™ Renal Denervation System (Experimental): Following angiogram, subjects found anatomically eligible and randomized to the renal denervation arm will be treated with the TIVUS™ Renal Denervation System.
  Interventions: Device: TIVUS™ Renal Denervation System
- Sham (Sham Comparator): For those subjects randomized to the sham control, the angiogram will serve as the sham procedure.
  Interventions: Other: Sham

INTERVENTIONS:
Device: TIVUS™ Renal Denervation System — Renal artery catheterization procedure used to denervate the renal sympathetic nerves in the perivascular space using ultrasound energy.
  Other Names: Renal Denervation
  Arms: TIVUS™ Renal Denervation System
Other: Sham — For those subjects randomized to the sham control, the angiogram will serve as the sham procedure.
  Arms: Sham

SUMMARY:
The primary objective of the THRIVE Pivotal study is to demonstrate the adjunctive effectiveness and the safety of the TIVUS system in:

1. subjects with hypertension (HTN) receiving up to 2 anti-hypertensive drugs of different classes in whom the anti-hypertensive medications will be stopped for a 4-week wash-out period before RDN/Sham procedure and during 2 months after procedure.
2. subjects with controlled hypertension receiving up to 2 anti-hypertensive drugs of different classes and who accept to be off-medications for a 4-week wash-out period before RDN/Sham procedure and 2 months after the procedure

DETAILED DESCRIPTION:
THRIVE is an international, multicenter, randomized, double blind, sham-controlled study, designed to demonstrate the adjunctive effectiveness and safety of the TIVUS System in hypertensive subjects while subjects are maintained off-antihypertensive medications for a 4-week wash-out period before RDN/Sham procedure and 2 months after procedure. At two months after procedure, subjects with uncontrolled hypertension are put back on antihypertensive medication according to a medication escalation protocol. Unblinding will be performed at 6 months. Uncontrolled sham subjects can cross-over to RDN procedure at 6-months. The sham procedure will be minimally invasive to reduce risk to subjects. All subjects treated with TIVUS will be followed for a maximum of 36 months post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Appropriately signed and dated informed consent
2. Male and female adults with age between ≥22 and ≤75 years at time of consent
3. Documented history of hypertension
4. Previously or currently prescribed antihypertensive therapy
5. Subject has an office BP (average of 3 seated measurements) of:

   1. Uncontrolled BP: ≥ 140/90 mmHg <180/110 mmHg at Screening Visit (V0) while stable for at least 4 weeks on 0-2 anti-hypertensive medications of different classes* and willing to stop anti-hypertensive medication(s) for 4 weeks wash-out and 2-months post-procedure, (subjects with a history of treatment with anti-hypertensive medications but are not currently taking any at screening will undergo a 4-week run-in period) or,
   2. Controlled BP: < 140/90 mmHg while stable for at least 4 weeks on 1-2 antihypertensive medications of different classes and willing to stop anti-hypertensive medication(s) for 4 weeks wash-out and 2-months post-procedure
6. Able and willing to comply with all study procedures
7. Subject is willing to have and is a good candidate for conscious sedation

Subjects who meet the following criteria will be considered eligible for randomization:

* Documented daytime systolic ABP ≥ 135 mmHg and < 180 mmHg after 4-week washout/run-in period.**
* Suitable renal anatomy compatible with the renal denervation procedure, documented by renal CTA or MRA of good quality performed within one year prior to consent (a CTA or MRA will be obtained in subjects without a recent (≤1 year) cross-sectional renal imaging). The renal angiogram procedure done in the cath lab prior to randomization will serve as the final anatomy compatibility check.

  * Potassium-sparing diuretics such as Amiloride hydrochloride and Triamterene may be prescribed in combination with another diuretic (e.g. a thiazide or loop diuretic) for their potassium conservation properties. In this situation, the diuretic combination is considered as a single class of anti-hypertensive.

Exclusion Criteria:

1. Subject has been previously diagnosed with abnormal renal artery anatomy and/or renal anatomy such as a single kidney, ectopic or horseshoe kidney, polycystic kidney disease, kidney tumors or other findings precluding renal denervation therapy as detailed in the angiographic exclusion criteria
2. Uncorrected causes of secondary hypertension other than sleep apnea (including, but not limited to): aldosteronism, renal parenchymal disease, renovascular disease, excess catecholamines, Cushing's syndrome, erythropoietin use, pheochromocytoma, hypo/hyperthyroidism, hyperparathyroidism, acromegaly)
3. Type I diabetes mellitus or uncontrolled Type II diabetes (defined as a plasma HbA1c ≥ 9.0%)
4. eGFR of <40 mL/min/1.73 m2 CKD-EPI as calculated using the CKD-EPI 2021 equation
5. Cerebrovascular event (e.g. stroke, transient ischemic event, cerebrovascular accident) within 6 months prior to consent
6. History of severe cardiovascular event (e.g. myocardial infarction, unstable angina, CABG, acute heart failure requiring hospitalization (NYHA III-IV) within 12 months prior to consent
7. Subject has severe valvular stenosis or insufficiency
8. Documented repeat (>1) hospitalization for hypertensive crisis within the prior 12 months and/or any hospitalization for hypertensive crisis within three (3) months prior to consent
9. Prescribed to any standard antihypertensive cardiovascular medication (e.g. beta blockers) for other chronic conditions (e.g. ischemic heart disease) such that discontinuation might pose serious risk to health in the opinion of the investigator
10. Subject with rapid, uncontrolled, symptomatic atrial fibrillation
11. Active implantable medical device (e.g. ICD or CRT-D; neuromodulator/spinal stimulator; baroreflex stimulator)
12. Chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea.
13. Subject has a planned major surgery (any procedure requiring general anesthesia) in the next 12 months.
14. Subject on anticoagulant therapy that cannot be temporarily withheld for study procedure.
15. Primary pulmonary hypertension
16. Documented contraindication or allergy to contrast medium not amenable to treatment
17. Limited life expectancy of < 1 year at the discretion of the Investigator
18. Night shift worker
19. Subject has frequent intermittent or chronic pain that results in treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) for two or more days per week over the month prior to enrollment.
20. Subject is taking immunosuppressive therapy for diseases featuring vasculitis
21. Any known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or for any reason in the opinion of the investigator, would be unlikely or unable to comply with study protocol requirements or whose participation may result in data analysis confounders
22. Pregnant, nursing or planning to become pregnant within 12 months post procedure.

    Negative pregnancy test required, documented within a maximum of 7 days prior to procedure for all women of childbearing potential. Documentation of effective contraception is also required for women of childbearing potential
23. Subject has a planned major surgery or cardiovascular intervention in the next 6 months
24. Subject with history of renal transplantation
25. Evidence of active infection within 7 days of procedure (based on positive lab test and requiring therapy).
26. Subject has hypertrophic cardiomyopathy or amyloidosis.
27. Prior renal denervation procedure
28. Concurrent enrollment in any other investigational drug or device trial (participation in non-interventional studies/registries is acceptable)
29. Subject on a beta blocker for a condition other than antihypertension

Angiographic Exclusion Criteria:

The following characteristics identified either on the renal artery CT scan or MRI or on the Eligibility II Renal artery Angiogram will prevent the subject from being included:

1. Main renal arteries lumen diameter < 4 mm.
2. Main renal treatable artery length <20mm (may include proximal branching).
3. Accessory renal arteries that supplies ≥ 25% of the parenchyma, and < 4 mm in lumen diameter.
4. Aorto-renal angle that prevents a safe cannulation of the renal artery.
5. Severe common femoral artery, common and/or external iliac artery, renal, iliac or aortic calcification or tortuosity that may compromise the safe performance and completion of the TIVUS™ procedure.
6. Hemodynamically or anatomically significant renal artery abnormality or stenosis in either renal artery which, would interfere with safe cannulation of the renal artery or meets local standards for surgical repair or interventional dilation (NOTE: vessel areas with calcification and fibromuscular dysplasia (FMD) should be avoided as intended treatment areas).
7. Any renal artery stenosis > 30% by visual assessment.
8. Any renal artery aneurysm (>50% of the main renal artery reference vessel diameter by visual estimate).
9. Presence of fibromuscular dysplasia of the renal arteries
10. Significant renal artery atheroma, aneurysm, calcification in the target vessel identified on CT Angiogram

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2028-08-15 (Estimated)

PRIMARY OUTCOMES:
Reduction in average daytime ambulatory systolic BP | From baseline to 2 months post-procedure
  Primary outcome
Subject level composite of the incidence of Major Adverse Events (MAE) | From Baseline to 30 day and 6 months post procedure
  Safety outcome

SECONDARY OUTCOMES:
Reduction in average 24-hr ambulatory systolic BP | From baseline to 2 Months post procedure
  Secondary outcome
Reduction in average home systolic BP | From baseline to 2 Months post procedure
  Secondary outcome
Reduction in average office systolic BP | From baseline to 2 Months post procedure
  Secondary outcome
Reduction in average daytime ambulatory diastolic BP | From baseline to 2 Months post procedure
  Secondary outcome
Reduction in average 24-hr ambulatory diastolic BP | From baseline to 2 Months post procedure
  Secondary outcome
Reduction in average home diastolic BP | From baseline to 2 Months post procedure
  Secondary outcome
Reduction in average office diastolic BP | From baseline to 2 Months post procedure
  Secondary outcome
Percentage of subjects with Systolic Blood Pressure (SBP) at target (daytime SBP <135 mmHg; office SBP <140 | From baseline to 2 and 6 Months post procedure
  Secondary outcome
Percentage of subjects with SBP at target (daytime SBP <135 mmHg; office SBP <140 mmHg) in the absence of. changes in hypertensive medication in each arm | From baseline to 2 and 6 Months post procedure
  Secondary outcome
Incidence of ambulatory systolic BP (daytime/24-hr/night-time) reductions of ≥5 mmHg, ≥10 mmHg, and ≥15 mm Hg | From baseline to 2, 6, and 12 Months post procedure
  Secondary outcome

OTHER OUTCOMES:
Reduction in average night-time ambulatory systolic/diastolic BP | From baseline to 2, 6 and 12, Months post procedure
  Observational outcome
Reduction in average daytime & 24-hr ambulatory systolic BP at 6- and 12-months post procedure. | From baseline to 6 and 12 Months post procedure
  Observational outcome
Reduction in average daytime & 24-hr ambulatory diastolic BP | From baseline to 6 and 12 Months post procedure
  Observational outcome
Reduction in average office systolic BP | From baseline to 6 and 12 Months post procedure
  Observational outcome
Reduction in average home systolic/diastolic BP | From baseline to 1, 3, 4, 5, 6, and 12-Months post procedure
  Observational outcome
Reduction in office and ambulatory pulse pressure | From baseline to 2, 6 and 12 Months post procedure
  Observational outcome
Reduction in office and ambulatory heart rate | From baseline to 2, 6, and 12 Months post procedure
  Observational outcome
Antihypertensive medication burden (number of antihypertensive drugs, doses, classes) | From baseline to 2, 6 and 12 Months post procedure
  Observational outcome
Percentage of subjects meeting escape criteria | From baseline to 2 Months post procedure
  Observational outcome
Percentage of subjects requiring initiation of antihypertensive drug therapy | From baseline to 2 and 6 Months post procedure
  Observational outcome
Percentage of subjects without any antihypertensive treatment | From baseline to 6 and 12 Months post procedure
  Observational outcome
Percentage of subjects requiring initiation of anti-hypertensive drug therapy at any available time points post procedure | From baseline through completion of study
  Observational outcome
Change in adherence to medications assessed by urine chemical adherence testing using liquid chromatography with tandem mass spectrometry (LCMSMS) | From baseline to 2, 6, 12, 24 and 36 Months.
  Observational outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Kirtane, MD, Study Chair — Columbia University; Michel Azizi, MD, Study Chair — George Pompidou Hospital; Felix Mahfoud, MD, Study Chair — University of Basel
Locations (44):
- United States (30):
  - Cardiology, PC, Birmingham, Alabama
  - Honor Health Research Institue, Scottsdale, Arizona
  - St. Bernard's Medical Center, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Cedar-Sinai Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - Bridgeport, Bridgeport, Connecticut
  - Ascension- Sacred Heart, Pensecola, Florida
  - University of South Florida, Tampa, Florida
  - Ascension Alexian Brothers, Elk Grove Village, Illinois
  - St. John's Prairie Heart, Springfield, Illinois
  - Southern Illinois University, School of Medicine, Springfield, Illinois
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Providence Hospital, Southfield, Michigan
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Jackson Heart, Jackson, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - St Lukes Hospital, Kansas City, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - Virtua Health, Camden, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Nyph/Cumc, New York, New York
  - NC Heart and Vascular, Raleigh, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical City, Fort Worth, Texas
  - Houston Medical Center, Houston, Texas
  - St Marks Hospital, Salt Lake City, Utah
  - Chippenham Hospital, Richmond, Virginia
- France (2):
  - Hopital Saint André, Bordeaux
  - Hôpital Européen Georges-Pompidou, Paris
- Germany (7):
  - Universitätsklinikum Erlangen, Erlangen
  - Frankfurt Sankt Katharinen Krankenhaus, Frankfurt
  - Freiburg Herzzenrtum, Freiburg im Breisgau
  - Marienkrankenhaus Hamburg, Hamburg
  - Herne Marien Hospital, Herne
  - Herzzentrum Leipzig, Leipzig
  - Sana Kliniken Lubeck, Lübeck
- Greece (3):
  - Athens Hippokration, Athens
  - University of Crete, Heraklion
  - Thessaloniki Hippokration General Hospital, Thessaloniki
- Italy (2):
  - Clinica Montevergine, Mercogliano
  - Ospedale Sant'Andrea, Roma

IPD SHARING:
Plan to Share IPD: No